CLINICAL TRIAL: NCT04887493
Title: Efficacy and Safety of Sublingual Versus Vaginal Misoprostol for Induction of Labor for Primigravida at 41 or More Weeks of Pregnancy: A Randomized Clinical Trial
Brief Title: To Study the Efficacy and Safety of Misoprostol by Sublingual Routes for Induction of Labour
Acronym: SL-IOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Bhutan (Other Government)
Responsible Party: Principal Investigator, Yeshey Dorjey, Principal Investigator, Ministry of Health, Bhutan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sublingual misoprostol; IOL (Other: Phuentsholing Hospital, Chukha, Bhutan)
Record Dates: First submitted 2021-05-04; First posted 2021-05-14 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Induction of Labour
Keywords: Induction of labour; Sublingual misoprostol; Vaginal misoprostol; Vaginal delivery
MeSH Terms: interventions — Misoprostol; Alprostadil

STUDY DESIGN:
Intervention Model Description: Pregnant mothers at term (37 - 42 weeks of gestation) and post term (>42 weeks of gestation) admitted to gynecology ward for induction of labour will be recruited to the study. The enrolled pregnant mothers will be randomly assigned to two groups by lottery method. Group 1- will be receive misoprostol 25µg by sublingual route for induction of labour; Group 2- will receive misoprostol 25µg by per vaginal route.
Who Masked: Outcomes Assessor
Masking Description: The participants and the investigators will not be masked; however, outcome assessor (statisticians) will be masked because they will not know anything about the drugs received by sublingual or per vaginal routes as their role will be to analyze the outcome only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sublingual misoprostol (Experimental): Sublingual misoprostol group will receive misoprostol 25µg by sublingual routes; the dose will be given repeatedly every 4 hours by sublingual route till there is labour pain or contraction or to a maximum of 6 dosages.
  Interventions: Drug: Misoprostol
- Vaginal misoprostol (Experimental): Vaginal misoprostol group will receive misoprostol 25µg by per vaginal routes; the dose will be given repeatedly every 4 hours by per vaginal route till there is labour pain or contraction or to a maximum of 6 dosages.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Misoprostol 25µg will be used for both the study arms
  Other Names: Prostaglandin E1

SUMMARY:
This research is to compare the efficacy and the safety of sublingual misoprostol with vaginal misoprostol administration for the induction of labour for primigravida at 41 or more weeks of pregnancy. In routine practice, misoprostol 25µg is used by per vaginal route for the induction of labour in Bhutan. The misoprostol dose is given repeatedly every 4 hours to a maximum of 6 dosages. The per vaginal route is found to be very effective and safe for the induction of labour. But, patient compliance is poor and increasing the risk of neonatal sepsis since it has to be inserted into vagina every 4 hours. To overcome these problems with per vaginal route, this study is developed to explore the efficacy and safety of misoprostol use by sublingual routes for the induction of labour. Misoprostol can be used by sublingual, oral or per vaginal route as per the findings of the other studies.

If the finding of this study proves sublingual use of misoprostol is safe and efficient for the induction of labour, the current practice of using misoprostol by vaginal route will be changed to sublingual route in Bhutan.

DETAILED DESCRIPTION:
Induction of labour is an intervention intended to artificially initiate uterine contraction in pregnant women who are not in labour. It is a common practice to interrupt the pregnancy at 41 weeks of gestation and deliver the fetus when continuation of pregnancy is no longer considered safe.

The methods of induction can be non-pharmacological or pharmacological. Prostaglandins and oxytocin are the commonly used drugs for induction of labour.

Prostaglandins are the current drug of choice and have been used for labour induction in pregnant women with an unfavourable cervix. Misoprostol is a synthetic analogue of prostaglandin E1 and it has been extensively and successfully used for labour induction due to its efficacy, low cost and stability at room temperature. Misoprostol can be used by oral, vaginal or sublingual routes for the labour induction. Among which vaginal misoprostol has been extensively used and shown to be an effective method of induction of labour. Sublingual route of misoprostol is equally safe and effective for induction of labour. In fact, sublingual route of misoprostol administration is found to be more effective in induction of labour as compared to vaginal route. This sublingual route is appealing for several reasons, including the convenience, easy to administer and a higher patient's acceptability. In contrast to per vaginal misoprostol administration, sublingual route avoids repeated per vaginal examination which is a risk factor for neonatal sepsis.

In Bhutan per vaginal misoprostol is being extensively used for induction of labour by the Gynecologists. The neonatal sepsis rate is 19 per 1000 in Bhutan, which is the highest in Asia. The high rate of neonatal sepsis in Bhutan is found to be associated with repeated vaginal examination done during pregnancy to administer misoprostol dose.

No study has been conducted in Bhutan to find out the safety and efficacy of per vaginal misoprostol use nor is there any study on sublingual use of misoprostol for the induction of labour.

Therefore, this study is developed to explore whether sublingual misoprostol may be tried as a new option for induction of labour comparing the efficacy of administration of sublingual misoprostol with vaginal misoprostol for induction of labour at term and post term pregnancies.

This will be a randomized clinical trial with a parallel design (simple randomization).

The study will be conducted in Phuentsholing General Hospital, Chukha, Bhutan.

The study duration will be six months starting from 1st June to 30th November 2021.

For the study, all the primigravida at 41 or more weeks of pregnancy admitted to Gynecology ward, Phuentsholing hospital will be approached to participate.

Primigravid pregnant women who have consented voluntarily will be recruited for the study. The study population will randomly put into two groups by simple randomization as follows:

Group 1- To induce the labor with misoprostol 25µg sublingually; Group 2- To induce the labor with misoprostol 25µg per vaginally.

The researchers and the study participants will not be blinded; however, the statisticians who will analyze the data will be blinded to avoid possible bias in drawing the inferences.

Sample size is calculated based on the finding of previous study which had reported with a statistically significant difference of mean induction to delivery interval between sublingual group and per vaginal use of misoprostol group (P<0.001). The mean induction to delivery interval of 13.1±4.1 hours for sublingual group as compared to 17.9±5.4 hours for vaginal group(21). With 5% error and 80% power, sample size is determined by using PASS (Power Analysis and Sample Size Software) 2021 software.

The total sample size is 24 from the calculation using the previous research finding.

Therefore, the current research will recruit 20 study participants in each group; group 1 (n=20), and group 2 (n=20).

Sampling technique will be a non-purposive sampling.

Written informed consent will be obtained from the participants.

After obtaining ethical clearance from the Research Ethical Board of Health (REBH), Ministry of Health, Thimphu, Bhutan; pregnant women who are admitted to gynecology ward for induction of labor for various reasons will be approached and will take detailed history, review previous medical documents, and conduct relevant general and obstetrical examination. This procedure will be done to ensure correct dating of pregnancy (to avoid inducing preterm), to re-confirm the indications for induction of labor and to exclude contraindications for vaginal delivery. Primigravid pregnant women at 41 or more weeks of pregnancy will be counseled and explained about the research purpose, objectives, methods, outcomes and the benefits. If they are willing to participate in the research, the written informed consent will be obtained. Eligibility criteria will be applied and the pregnant mothers who fulfill the inclusion criteria will be recruited for the study from 1st June to 30th November 2021.

The enrolled pregnant women will then be randomly allocated in two groups by lottery methods. Enrolled pregnant mothers will be asked to pick up a rolled paper from the lottery box which will determine the study group of the subject. The group-1 will receives misoprostol 25µg by sublingual route and group-2 will receives misoprostol 25µg by vaginal route. Sublingual route involves placing misoprostol in the sublingual space under the tongue and the vaginal route involves placing misoprostol inside the posterior fornix of vagina.

Prior to starting the first dose of misoprostol administration, cardiotocography (CTG) will be done to ensure fetal heart rate tracing is reassuring and per vaginal examination will be done to assess the Bishop's score in both the groups.

Per vaginal examination will be done by a female nurse maintaining optimum privacy. If the fetal heart rate is reassuring and the Bishop's score is unfavorable, then induction of labor with misoprostol will commence. Both groups will receive repeat dose of misoprostol 25µg every 4 hours up to a maximum of 6 dosages. The drug will be administered sublingually or vaginally according to the allocated group by the female nurse.

Pregnant women will never be left unattended once the induction of labor has started. Close monitoring of fetal heart rate and uterine activity will be done for 30 minutes after every dose of misoprostol for both the study group. This is to look for changes in fetal heart rate and for early detection of rare occurrence of uterine hyperstimulation with the peak concentration of misoprostol in the circulation. If there is uterine hyperstimulation (presence of five or more contractions per 10 minutes for at least 20 minutes) patient will be monitored with continuous CTG, put patient on left lateral position, give oxygen (8-10L/min) and hydrate with IV fluids. If hyperstimulation fails to resolve and the abnormal fetal heart rate persists (absence of acceleration, presence of late or variable deceleration, reduced variability, bradycardia or tachycardia) Inj. salbutamol 100 µg IV over 1-2 minute will be given. If CTG remains suggestive of fetal compromise despite the management for hyperstimulation, pregnancy will be terminated by emergency caesarean section.

Prior to repeating the misoprostol dose, repeat CTG will be done to ensure reassuring fetal heart rate tracing in both the groups. For group 2 per vaginal examination will be done every 4 hours to assess Bishop score and to give a repeat dose of misoprostol per vaginal route. For group 1, repeated per vaginal examination will not be done, rather repeat misoprostol dose will be placed in the sublingual space under the tongue. The repeat misoprostol dose will be administered only if fetal heart rate tracing is reassuring and there is no uterine contraction or labor pain. If the fetal heart rate tracing is non-reassuring (fetal distress), the repeat dose of misoprostol will be withheld and pregnant mothers will be put to left lateral position, IV fluids (crystalloids) will be given to hydrate, oxygen will be administered by face mask at 6-10L/min and CTG will be repeated after 30minutes. If the fetal heart rate tracing is still non-reassuring (features of fetal distress persists) even after managing with hydration and oxygen administration, pregnancy will be terminated by emergency caesarean section.

If fetal heart rate tracing returns to reassuring status after hydration and oxygenation, the misoprostol dose will be restarted. Once the uterine contraction or labor pain starts, the repeat dose of misoprostol will be withheld and per vaginal examination will be done for both the study groups to assess the Bishop score. Once the cervix becomes ripe or the Bishop score is favorable, and in absence of uterine contraction or labour pain, induction with oxytocin will be done after 4 hours of the last dose of misoprostol administration.

Once the patient is in active labor, augmentation with oxytocin will be done if there is inadequate uterine contraction. Labor process will be closely monitored for progression of labor and to assess fetal and maternal conditions using partograph. Routine active management of the third stage of labor will be done.

Newborn will be assessed for Apgar score at 1 minute and again at 5 minutes after birth.

In both the study groups if labor fails to get induced even after 6 dosages of misoprostol (failed induction), and if Bishop score is unfavorable; induction with Foley's catheter will be offered to the pregnant mother. Foley's catheter (16F) will be placed by transcervically and inflate the balloon with 30-50 ml of water. Unless balloon expels out it is kept in situ for 12 hours. After 12 hours Foley's catheter will be removed by deflating the balloon. If the labour fails to get induced or the Bishop score is unfavorable even after the mechanical induction with Foley's catheter, pregnancy will be terminated by caesarean section.

After the delivering the baby, and when mothers are free of pain, they will be asked to give a rating on the satisfaction score scale on the induction of labour route they received.

The interviewer administered pre-tested questionnaire will be used to collect the data. Pre-testing of the questionnaire will be done to the gynecology ward nursing staff.

Primary outcome is to measure the number of pregnant mothers who have a vaginal delivery within 24 hours of the induction.

Secondary outcomes are; to find out the time taken from induction to delivery, to find out the total dosages of misoprostol required for induction, to find out the maternal and neonatal outcomes, to measure the satisfaction score and to analyze the Apgar score at birth.

The study proposal is submitted to the Research Ethical Board of Health (REBH), Ministry of Health, Thimphu, for ethical clearance and an expedited review. The research will commence only after obtaining ethical clearance.

The collected data will be captured and double entered using Epidata 3.1.2 (Odense, Denmark) and validated to avoid data entry errors. The data will then be exported to SPSS format for further analysis. The data will be analyzed using SPSS version 23. Descriptive statistics commands such as frequencies, percentages, mean, median, confidence interval, and standard deviation will be used to describe the study variables. The Chi-square test will be used for categorical variables outcome variables. Student's t-test will be employed for A p value <0.05 will be considered statistically significant with confidence interval of 95%.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more years
* Primigravida
* Singleton pregnancy
* Gestation at 41 or more weeks of pregnancy
* Estimated fetal weight of <4000 gram
* In cephalic presentation
* Bishop score < 6 (unfavorable cervix)
* Reassuring fetal heart rate tracing

Exclusion Criteria:

* Age <18 years
* Multiple pregnancy (twin, triplet and higher order pregnancies)
* Gestation <41 weeks of pregnancy
* Fetal macrosomia (Estimated fetal weight >4000 gram)
* Cephalo-pelvic disproportion
* Malpresentation (breech, oblique, transverse)
* Bishop score >6 (favorable cervix)
* Presence of labor or uterine contractions
* Non-reassuring fetal heart rate tracing
* Pregnant women with known allergy to misoprostol,
* Previous Caesarean delivery or other uterine surgery
* Previous uterine rupture
* Placenta previa
* Chorioamnionitis
* Prelabour rupture of membrane (PROM)
* Antepartum hemorrhage (per vaginal bleeding)
* Contraindication to vaginal birth
* Medical disorders in pregnancy
* Active genital herpes infection
* Invasive cervical carcinoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The person with female gender gets pregnant. A male person is not compatible to get pregnant. The study will recruit only those pregnant mothers who need induction of labour.
Enrollment: 500 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
To measure the number of pregnant mothers who have a vaginal delivery within 24 hours of the induction. | The numbers of successful vaginal delivery conducted in each group will be measured for 6 months.
  The number of successful vaginal deliveries will be recorded and compared between the study arms. This is to study the overall efficacy of sublingual use of misoprostol in compared between the study group

SECONDARY OUTCOMES:
To compare the dosages of misoprostol required for induction of labour in the study arms. | The total number of repeat dosages of misoprostol use in the each study participant will be determined for 24 hours.
  The total dosages of misoprostol required to induce the labour will be recorded for both the study arms. The comparison will be done to see which study arm required maximum repeat dosages of misoprostol for induction of labour.
The modes of delivery will be compared between the study arms | The individual modes of delivery will be documented for 24-48 hours
  The modes of delivery for each arm of study will be recorded. The total numbers of vaginal deliveries, instrumental vaginal deliveries, and total Caesarean section performed will be collected in the data collection sheet. The collected data will be analyzed to see which study arm has more vaginal deliveries as compared to Caesarean delivery. The study arm which has more vaginal deliveries will be considered as more efficient and safe as compared to other arm.
To compare the induction to delivery interval between the study group | The time taken from the starting of the induction to the time at delivery will be measured for individual study participant for 24 - 48 hours.
  The time taken from the induction to vaginal delivery will be recorded and will be compared between the study group

CONTACTS AND LOCATIONS:
Overall Officials: Yeshey Dorjey, Principal Investigator — Ministry of Health, Phuentsholing Hospital, Chukha, Bhutan
Locations (1):
- Phuentsholing Hospital, Phuentsholing, Bhutan

IPD SHARING:
Plan to Share IPD: No
I will decide later and provide updates here

REFERENCES:
- [Background] Teixeira C, Lunet N, Rodrigues T, Barros H. The Bishop Score as a determinant of labour induction success: a systematic review and meta-analysis. Arch Gynecol Obstet. 2012 Sep;286(3):739-53. doi: 10.1007/s00404-012-2341-3. Epub 2012 May 1. PMID 22546948
- [Background] Batinelli L, Serafini A, Nante N, Petraglia F, Severi FM, Messina G. Induction of labour: clinical predictive factors for success and failure. J Obstet Gynaecol. 2018 Apr;38(3):352-358. doi: 10.1080/01443615.2017.1361388. Epub 2017 Oct 23. PMID 29058493
- [Background] Mozurkewich EL, Chilimigras JL, Berman DR, Perni UC, Romero VC, King VJ, Keeton KL. Methods of induction of labour: a systematic review. BMC Pregnancy Childbirth. 2011 Oct 27;11:84. doi: 10.1186/1471-2393-11-84. PMID 22032440
- Available data/document: Study Protocol: Misoprostol — https://www.researchgate.net/publication/351331713_Efficacy_and_Safety_of_Sublingual_versus_Vaginal_Misoprostol_for_Induction_of_Labor_at_Term_and_Post_Term_Pregnancies_A_Randomized_Clinical_Trial_Efficacy_and_Safety_of_Sublingual_versus_Vaginal_Misop